CLINICAL TRIAL: NCT04560699
Title: Targeted Physiotherapeutic Treatment for Aromatase Inhibitor-associated Musculoskeletal Pain in Breast Cancer Survivors: a Randomized Controlled Trial
Brief Title: Targeted Physiotherapeutic Treatment for Aromatase Inhibitor-associated Musculoskeletal Pain in Breast Cancer Survivors
Acronym: AIMSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Cecilie Bartholdy, Principal investigator, Frederiksberg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APPI2-PT-2020-AIMSS
Record Dates: First submitted 2020-09-16; First posted 2020-09-23 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Musculoskeletal Pain
Keywords: aromatase inhibitors; breastcancer survivors
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: randomized 1:1 to intervention or control
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator is masked to group assignment for study analysis. Outcome assessor is masked to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapeutic group (Active Comparator): medical care and physiotherapeutic treatment
  Interventions: Other: Physiotherapeutic treatment and medical care
- medical care group (Active Comparator): Medical care
  Interventions: Other: medical care

INTERVENTIONS:
Other: Physiotherapeutic treatment and medical care — Physiotherapeutic treatment twice a week for twelve weeks and medical care three times at baseline, week 13 and week 26
  Arms: Physiotherapeutic group
Other: medical care — medical care three times during the study period; baseline, week 13 and week 26
  Arms: medical care group

SUMMARY:
The primary objective of this trial is to assess the efficacy of targeted individualised physiotherapeutic treatment on aromatase inhibitor-associated musculoskeletal pain.

This trial asks a critical, previously unaddressed, question of clinical importance about management of musculoskeletal (MSK) pain secondary to aromatase inhibitor (AI) treatment of hormone receptor-positive breast cancer. Many breast cancer survivors taking AIs experience muscle and/or joint pain, which may cause many to stop taking AIs and may inhibit exercise or physical activity, despite its known health benefits.

Physiotherapeutic treatment is considered a standard management strategy for many MSK pain conditions, in which targeted specific exercise therapy is now as an evidence-based management strategy with proven effectiveness and patient satisfaction. Thus, referral to physiotherapy would be a natural strategy in women who experience MSK pain as an adverse effect to AI therapy. However, it is unclear if physiotherapeutic treatment has similar effects on AI induced MSK pain as in primary MSK pain. Two systematic review (one with a meta-analysis) have assessed the effect of different pain management strategies for AI-induced MSK-pain and found great uncertainty in the effects of exercise, relaxation techniques and acupuncture. They also found limited evidence on the subject and moderate to low quality of the studies included. The evidence on the subject is clearly limited but the need for a treatment option to minimize the side-effects of the AI medication real and necessary.

Targeted individualised physiotherapeutic treatment is tailored for the affected (painful) tissue/joint/region specifically and is based on extensive experience and evidence from MSK physiotherapy in rheumatic and orthopedic patient population. Targeted individualised physiotherapy treatment take into account the individual patient, her constitution, the painful tissue/region/joint (e.g. its biomechanics, physiological properties, and inflammatory activity), and is adjusted according to day-to-day variations in pain and progressed based on the interaction between changes in symptoms and function and tissue healing. Such approach is expected to yield a greater effect on MSK pain, than a generic exercise program. Further, targeted treatment programs are delivered by trained physiotherapists, who have specific clinical training and experience in clinical management of patient and handling MSK pain, which is also expected to yield better clinical outcomes than programs delivered by people without clinical training.

Altogether it is very likely that a targeted physiotherapy treatment will be of significant benefit to breast cancer survivors with AI induced MSK pain.

The aim is to compare targeted individualized physiotherapeutic treatment and medical care with medical care alone on aromatase inhibitor associated musculoskeletal pain in female breast cancer survivors.

It is hypothesized that targeted physiotherapeutic treatment and medical care reduces musculoskeletal pain significantly in women with aromatase inhibitor associated musculoskeletal pain when compared to medical care alone.

The plan is to include 120 participants from the oncology department at Rigshospitalet, Denmark.

Participants will partake in the study for a total of 26 weeks. During the first 12 week the intervention group will receive the physiotherapeutic treatment twice a week. The medical care visits are place at the first visit to the clinic, week 13 and week 26.

DETAILED DESCRIPTION:
The primary objective of this trial is to assess the efficacy of targeted individualised physiotherapeutic treatment on aromatase inhibitor-associated musculoskeletal pain.

This trial asks a critical, previously unaddressed, question of clinical importance about management of musculoskeletal (MSK) pain secondary to aromatase inhibitor (AI) treatment of hormone receptor-positive breast cancer. Many breast cancer survivors taking AIs experience muscle and/or joint pain, which may cause many to stop taking AIs and may inhibit exercise or physical activity, despite its known health benefits.

Physiotherapeutic treatment is considered a standard management strategy for many MSK pain conditions, in which targeted specific exercise therapy is now as an evidence-based management strategy with proven effectiveness and patient satisfaction. Thus, referral to physiotherapy would be a natural strategy in women who experience MSK pain as an adverse effect to AI therapy. However, it is unclear if physiotherapeutic treatment has similar effects on AI induced MSK pain as in primary MSK pain. Two systematic review (one with a meta-analysis) have assessed the effect of different pain management strategies for AI-induced MSK-pain and found great uncertainty in the effects of exercise, relaxation techniques and acupuncture. They also found limited evidence on the subject and moderate to low quality of the studies included. The evidence on the subject is clearly limited but the need for a treatment option to minimize the side-effects of the AI medication real and necessary.

Targeted individualised physiotherapeutic treatment is tailored for the affected (painful) tissue/joint/region specifically and is based on extensive experience and evidence from MSK physiotherapy in rheumatic and orthopedic patient population. Targeted individualised physiotherapy treatment take into account the individual patient, her constitution, the painful tissue/region/joint (e.g. its biomechanics, physiological properties, and inflammatory activity), and is adjusted according to day-to-day variations in pain and progressed based on the interaction between changes in symptoms and function and tissue healing. Such approach is expected to yield a greater effect on MSK pain, than a generic exercise program. Further, targeted treatment programs are delivered by trained physiotherapists, who have specific clinical training and experience in clinical management of patient and handling MSK pain, which is also expected to yield better clinical outcomes than programs delivered by people without clinical training.

Altogether it is very likely that a targeted physiotherapy treatment will be of significant benefit to breast cancer survivors with AI induced MSK pain.

The aim is to compare targeted individualized physiotherapeutic treatment and medical care with medical care alone on aromatase inhibitor associated musculoskeletal pain in female breast cancer survivors.

It is hypothesized that targeted physiotherapeutic treatment and medical care reduces musculoskeletal pain significantly in women with aromatase inhibitor associated musculoskeletal pain when compared to medical care alone.

The plan is to include 120 participants from the oncology department at Rigshospitalet.

Participants will partake in the study for a total of 26 weeks. During the first 12 week the intervention group will receive the physiotherapeutic treatment twice a week. The medical care visits are place at the first visit to the clinic, week 13 and week 26.

Allocation of participants and sequence generation The randomization list will be computer-generated based upon permuted random blocks of variable size (4 to 6 in each block). The allocation ration will be 1:1 (1 targeted physiotherapeutic treatment (TPT)+ medical care (MC) for each 1 MC) stratified according to upper or lower MSK pain site.

The biostatistician or his delegate will develop the randomisation scheme for allocation subjects to the two treatment arms.

Investigators, study coordinators, clinical staff, study staff, and other personnel directly involved in the study, will be blinded to the group allocation.

Participants and staff involved in the physiotherapy treatment are not blinded to the group allocation. Information that could potentially unblind otherwise blinded staff will not be shared, and will be stored in facilities with limited access until the study is completed. Unblinding of blinded personnel does not preclude the related participants' continued participation in the study.

Attendance to the physiotherapy sessions and the medical doctor appointments will be recorded in the case report form (CRF).

The investigator and clinical staff will monitor each participant for evidence of adverse events (AEs) throughout the study. The investigator will assess and record any AE in detail including the date of onset, description, severity, duration and outcome, relationship of the AE to study treatment, and any action(s) taken. AEs, whether in response to a query, observed by site personnel, or reported spontaneously by the participant will be recorded.

A participant may withdraw from the study at any time without this impacting on any future investigations and/or treatments at the site, by the Investigators in this study or by other staff associated with the study.

If a participant withdraws from the study, the procedures outlined for the closest assessment visit is sought to be completed within 2 weeks, and preferably prior to the initiation of another therapy. However, these procedures should not interfere with the initiation of any new treatments or therapeutic modalities that the investigator feels are necessary to treat the participant's condition.

All AEs will be followed to a satisfactory conclusion. The investigator may discontinue any participant's participation for any reason, including an AE, safety concerns or failure to comply with the protocol.

Participants will be discontinued from the study immediately if any of the following occur:

* Clinically significant abnormal laboratory results or AEs, which rule out continuation of the study treatment, as determined by the investigator
* Death
* Other illness
* Failure to adhere to the protocol

If at any point in time between randomization and the week-26 visit the investigator feels that the patient's clinical course is not acceptable within the normally applied paradigms of AIMSS, the patient should be taken out of the study. The clinician's judgment will be required to decide on a case-by-case basis whether to implement this step or not.

It is important to avoid any loss to follow-up participants for the efficacy assessment and meaningful analysis of the study.

The principal investigator has the right to terminate this study at any time. Reasons may include the following, but are not restricted to:

* The incidence of events in this or other studies that indicate a potential health hazard to participants.
* Unsatisfactory participant enrolment. Determination of Sample Size This is a superiority study with the main outcome being change in pain from baseline to end of study (week 13), measured with the BPI.

Given a standard deviation of 2.5 a total sample size of 100 is required to obtain a power of 0.85 (actual power is 0.887) to detect a mean group difference in the change from baseline of 1.5 points at a significance level of 0.05 and using a balanced design (1:1 randomization). Allowing for drop-outs the study aims at recruiting and randomize 120 participants, which would yield a power of 0.935 to detect the above difference at the 0.05 level of significance.

Power and sample size analyses were conducted using 'SAS Power and Sample Size' (SAS Institute Inc., Cary, North Carolina).

Disposition of participants The number of randomized patients will be summarized as total using counts and percentages. The number of patients either completing or permanently discontinuing the study will be summarized using counts and percentages.

For the assessment of superiority, the intention-to-treat (ITT) protocol population is used in the primary analysis, as it is the most conservative approach.

The ITT population consist of all randomized patients irrespective of whether the patient actually received study intervention or the patient's compliance with the study protocol, in the treatment group to which the participant was assigned at randomisation. A patient will be considered randomised as soon as a treatment is assigned by according to the allocation sequence.

A statistical analysis plan that describes the details of the planned statistical analyses will be produced by the principal investigator and a biostatistician or his delegate before last patient's last visit.

Assessments of changes from baseline and construction of confidence intervals (CI) for continuous measures will be based on a repeated measures analysis of covariance (ANCOVA; including group as the main factor and baseline measure as covariate).

Superiority will be claimed if the computed 95% confidence interval of the estimated group difference in the change from baseline in the BPI does not include 0 in the ITT population.

All statistical tests will be two-sided and statistical significance will be claimed if the computed p-value is equal to or less than 0.05.

The study will use paper case report forms (CRF) and an in-house custom built electronic data capture system (Cirkeline) and REDCap (internet survey system for the 6-week assessment).

Paper based CRF allows for on the go registration of participation in the TPT + MC group as well as registration from the structured interview.

Cirkeline allows individual patients to supply questionnaire data at clinical visits via touch-screens in the clinic, as well as entering of study related data by the staff.

REDCap allows the participants to fill out the questionnaires from home via a secure web browser.

At the end of the trial, all data will be merged and stored in a database created by the Parker Institutes database manager.

The applications meet all regulatory standards and allow management of all activities related to clinical trials that ensures optimal resource use and safety according to good clinical practice and data protection legislation.

Regulatory Standards Participant confidentiality Participant medical information obtained by this study is confidential, and disclosure to third parties other than those noted below is prohibited.

With the participant's permission, medical information may be shared with his or her personal physician or with other medical personnel responsible for the participant's welfare.

If the data from this study are published, the presentation format will not include names, recognizable photos, personal information or other data which compromises the anonymity of participating participants.

The study will be conducted in accordance with the Data Protection Act and follow the General Data Protection Regulation. The study data management and data security procedures is approved by the Regional Knowledge Centre on Data Protection Compliance on behalf of the Danish Data Protection agency.

All data will be entered into a study database for analysis and reporting. Any data captured electronically will be stored electronically in a separate database according to standard procedures at The Parker Institute. Upon completion of data entry, the databases will be checked to ensure acceptable accuracy and completeness. System backups and record retention for the study data will be consistent with The Parker Institute standard procedures.

Individuals involved in study evaluations will be trained to perform the efficacy and safety evaluations described in the protocol.

The study has received funding from Danish Physiotherapists Association and The Oak Foundation (OCAY-13-309; covering running cost at the Parker Institute including this study), for the specific purpose to complete this study. None of the investigators have conflicts of interests related to the funding of this study. This information is disclosed to all participants in the written information material.

All sources of support (including technical and financial support) provided for this study is disclosed in the written information material and in publication of the study results. Funding is an ongoing process. All future financial and/or technical support to the study will be reported to the Danish health research ethical committee system and is disclosed to all participants (previous, current and potential).

The participants are insured by the Danish Patient Insurance Association.

ELIGIBILITY:
Inclusion Criteria:

* Adequately treated primary invasive breast cancer with surgery (breast conserving surgery or mastectomy) and radiotherapy if applicable
* Estrogen receptor positive tumor with staining of ≥10% tumorcells
* Aromatase inhibitor treatment
* Perceived musculoskeletal pain in the upper or lower extremities attributable to AI treatment for at least 2 month and a maximum of 24 months
* Age ≥18
* Willing and able to understand and participate in the study

Exclusion Criteria:

* Locally advanced breast cancer or distant metastases
* Lymphedema
* Inflammatory rheumatic diseases (rheumatoid arthritis, Psoriatic arthritis, etc.)
* Widespread or generalized pain syndrome (e.g. fibromyalgia)
* Lumbar or cervical nerve root compression
* Poly-arthrosis resulting in joint replacement surgery
* Any other condition or impairment that, in the opinion of the investigator, makes a potential participant unsuitable for participation or which obstruct participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Change in Brief pain inventory (BPI) | Change from baseline to week 13
  The BPI is a 14-item questionnaire developed for use in cancer patients, and assesses pain over the past week, reported on a 0-10 scale, where mild pain as a score of 3-4, moderate pain score of 5-7, and severe pain score of 8-10. The BPI consists of two subscales: pain severity and pain interference.

SECONDARY OUTCOMES:
Change in Health related quality of life | Change from baseline to week 13
  The European quality of life, five dimensions, 3 point Likert scale (EQ-5D-3L) questionnaire ( measures on a 3 point Likert scale; no problems, some problems, and extreme problems.
Adherence to aromatase-inhibitor (AI) drug | week 13
  participants are asked if the adhere to their AI-treatment
change in analgesics | change from baseline to week 13
  participants are asked if the take analgesics for their MSK pain
Activities of daily living questionnaire (ADL-Q) | baseline, week 6, week 13, week 26
  The ADL-Q was developed to measure perceived quality of different ADL activities. The ADL-Q consists of 12 domains and a total of 47 items: 31 Personal ADL (PADL) and 16 Instrumental ADL (IADL) items. The PADL items are rated within the last 24 hours and the IADL items are rated within the last week. Each item is rated with seven response categories reflecting independence, safety, efficiency, and effort/fatigue
Change in physical activity | change form baseline to week 13
  The questionnaire physical activity scale (PAS) is used to assess average activity level. The PAS consist of one question: how physically active are you during a regular day? Divide the 24 hours into relevant categories of activity: sleeping, sitting down watching tv/playing computer, low activity (for example doing laundry), moderate activity (for example cleaning), high intensity activity (for example running fast).
Change in Grip strength | change from baseline to week 13
  Grip strength will be measured using an electronic dynamometer (North Coast Medical Inc.). The maximal strength (in kilo gram) will be measured three times and the maximal value will be reported. Both the dominant and non-dominant hand will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Parker Instituttet, Frederiksberg Hospital, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
At the end of the study inclusion, it will be decided if any individual participant data will be made available to other researchers